CLINICAL TRIAL: NCT05257915
Title: A Real-world Clinical Study to Evaluate the Effectiveness and Safety of Perampanel as an add-on Treatment for Epileptic Seizure
Brief Title: A China RWS to Evaluate the Effectiveness and Safety of Perampanel as an add-on Treatment for Epileptic Seizure
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Beijing Children's Hospital (Other)
Responsible Party: Principal Investigator, Xiaodan Li, MD, Resident, Beijing Children's Hospital
Other Study IDs: BCHsjk-2020-Z-151
Record Dates: First submitted 2022-01-25; First posted 2022-02-25 (Actual); Last update posted 2022-02-25 (Actual); Status verified 2022-02

CONDITIONS: Epilepsy
Keywords: Epilepsy; Perampanel
MeSH Terms: conditions — Epilepsy | interventions — perampanel

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Perampanel: Epilepsy patients who had failed clinical treatment with 1-3 anti-epileptic drugs (AEDs) with the optimal dose and course of treatment and needed perampanel additional treatment.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — For patients ≥12 years old, the initial dose is 2 mg/d, and according to the clinical response and tolerance of the patient, the dose is increased to the minimum clinically effective dose in increments of 2 mg, and the interval between dose increases is not less than 2 weeks.
  For patients <12 years, according to the actual clinical situation, the initial dose and addition plan are judged by the investigator.
  Other Names: Fycompa

SUMMARY:
This study is a real-word clinical trial. The purpose of this study is to evaluate the effectiveness and safety of perampanel as an add-on treatment for epileptic seizure. The enrolled subjects were epilepsy patients who had failed clinical treatment with 1-3 anti-epileptic drugs (AEDs) with the optimal dose and course of treatment and needed additional treatment. The study was a real-world prospective clinical study, and the initial and maximum doses of perampanel were individualized by neurologists according to the patient's clinical situation.

DETAILED DESCRIPTION:
This is a multi-center, prospective, observational study. Subjects who meet all of the inclusion and none of the exclusion criteria will be received perampanel. Baseline seizure counts (frequency) data is collected by subjects or guardian/legally authorized representative, retrospectively.

It is expected to enroll 600 patients with epilepsy who are eligible for inclusion enrollment and receiving Perampenal from January 2021 to October 2021. The initial and maximum doses of perampanel were individualized by neurologists according to the patient's clinical situation. The patients were followed up for 6 months and recorded the frequency of seizures and self-assessment of improvement. Safety will be assessed by monitoring and recording of all of AEs and serious adverse events (SAEs), discontinuation during 6 months treatment (patient spontaneous reporting).

ELIGIBILITY:
Inclusion Criteria:

* Within 1 year before taking perampanel, the frequency of epileptic seizures was ≥1 time/month on average;
* 1-3 kinds of AEDs have been used, and the optimal dose and course of treatment have been reached, but the effect is not good. Perampanel is used as an additional treatment;
* Follow up for at least 3 months;
* Sign informed consent (if necessary).

Exclusion Criteria:

* Patients who have participated in other researches on antiepileptic drugs or medical devices;
* Inaccurate or unreliable clinical records according to the judgment of participating doctors;
* When the database is closed, the expected follow-up time is less than 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: epilepsy patients who had failed clinical treatment with 1-3 anti-epileptic drugs (AEDs) with the optimal dose and course of treatment and needed additional treatment.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
50% response rate of Perampanel | 6 months
  Proportion of subjects who have at least 50% reduction in total seizure frequency during the Maintenance Period relative to the Baseline

SECONDARY OUTCOMES:
Seizure-free rate of Perampanel | 6 months
  Proportion of subjects who achieve seizure-free status for total seizure during the Maintenance Period
Retention rate of Perampanel | 6 months
  Percentage of subjects still using perampanel after the Maintenance Period
Safety and Tolerability | 6 months
  Incidence of all of adverse events (AEs), serious adverse events (SAEs) and discontinuation from treatment

CONTACTS AND LOCATIONS:
Overall Officials: Fang Fang, Study Chair — Beijing Children's Hospital
Locations (5):
- China (5):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing TianTan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing University First Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University People's Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No